CLINICAL TRIAL: NCT00736476
Title: Phase I/II, Randomized, Observer-blind, Placebo-controlled, Single-Center Study of the Tolerability, Immunogenicity, and Efficacy of an Novartis' Investigational H. Pylori Vaccine in H. Pylori-Negative Adults
Brief Title: Efficacy and Safety of an H.Pylori Vaccine in H.Pylori-Negative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: V99P2; 2007-003511-31
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2016-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter pylori infection; vaccination; adults

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: H.pylori vaccines
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: H.pylori vaccines — 1 dose of H.pylori vaccine at 0, 1, and 2 months
  Arms: 1
Biological: Placebo Vaccine — Placebo Vaccine at 0, 1, and 2 months
  Arms: 2

SUMMARY:
To study the safety, immunogenicity and efficacy of an investigational H. pylori vaccine, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 - 40 years of age in good health
* HP uninfected
* not pregnant and agree to use birth control throughout the study (females who can become pregnant)

Exclusion Criteria:

* remote or current HP infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Otto von Guericke Universität Magdeburg, Magdeburg, Germany

REFERENCES:
- [Derived] Malfertheiner P, Selgrad M, Wex T, Romi B, Borgogni E, Spensieri F, Zedda L, Ruggiero P, Pancotto L, Censini S, Palla E, Kanesa-Thasan N, Scharschmidt B, Rappuoli R, Graham DY, Schiavetti F, Del Giudice G. Efficacy, immunogenicity, and safety of a parenteral vaccine against Helicobacter pylori in healthy volunteers challenged with a Cag-positive strain: a randomised, placebo-controlled phase 1/2 study. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):698-707. doi: 10.1016/S2468-1253(18)30125-0. Epub 2018 Jul 2. PMID 30042064
- [Derived] Nell S, Estibariz I, Krebes J, Bunk B, Graham DY, Overmann J, Song Y, Sproer C, Yang I, Wex T, Korlach J, Malfertheiner P, Suerbaum S. Genome and Methylome Variation in Helicobacter pylori With a cag Pathogenicity Island During Early Stages of Human Infection. Gastroenterology. 2018 Feb;154(3):612-623.e7. doi: 10.1053/j.gastro.2017.10.014. Epub 2017 Oct 21. PMID 29066327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single study center in Germany
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- Group I (HP Vaccine): Subjects received three injections of HP Vaccine at 0, 1, and 2 months, followed by H.pylori challenge(oral administration of infectious HP inoculum)1 month later.
- Group II (Placebo): Subjects received three injections of Placebo at 0, 1, and 2 months,followed by H.pylori challenge (oral administration of infectious HP inoculum)1 month later.
Period: Overall Study
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Started | 36 | 27
Completed | 35 | 27
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group I (HP Vaccine): Subjects received three injections of HP Vaccine at 0, 1, and 2 months.
- Group II (Placebo): Subjects received three injections of Placebo at 0, 1, and 2 months
- Total: Total of all reporting groups
Arm/Group | Group I (HP Vaccine) | Group II (Placebo) | Total
Number analyzed (Participants) | 36 | 27 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.7) | 24.0 (3.3) | 26.1 (5.1)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy (Defined as Prevention of Infection) of the HP Vaccine Compared to Placebo.
Description: The efficacy of the investigational vaccine to prevent infection following H.pylori challenge in healthy adults was determined in terms of percentage of subjects with positive HP infections in the vaccinated and unvaccinated groups(Placebo).
  Infection rates was assessed by invasive Upper Gastrointestinal Endoscopy (UGE)tests that included HP histopathology, HP culture and rapid urease test (RUT), and non-invasive HP tests which included urea breath test (UBT) and fecal antigen test (FAT).
Time Frame: 12 weeks post HP challenge
Population: Per-protocol dataset
Measure: Number; unit: Percentage of subjects
Groups:
- Group I (HP Vaccine): Subjects received three injections of H.pylori(HP) Vaccine at 0, 1, and 2 months, followed by a H.pylori challenge (oral administration of infectious HP inoculum) 1 month later.
- Group II (Placebo): Subjects received three injections of Placebo (only aluminum hydroxide adjuvant) at 0, 1, and 2 months, followed by a H.pylori challenge (oral administration of infectious HP inoculum) 1 month later.
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Number analyzed (Participants) | 14 | 13
Percentage of subjects
  UBT positive (non-invasive test) | 0 | 0
  FAT positive (non-invasive test) | 21 | 8
  HP culture positive (invasive test) | 36 | 46
  RUT positive (invasive test) | 7 | 0
  Histopathology positive (invasive test) | 7 | 0
  Positive HP infection (Invasive+non-invasive) | 36 | 46

2. Primary Outcome: Number of Subjects Reporting Solicited Local* and Systemic Adverse Events Following Vaccination
Description: To assess the tolerability of an HP vaccine versus placebo in terms of number of subjects reporting solicited local* and systemic adverse events.
Time Frame: Day 1-7 post vaccination
Population: This analysis was done on the safety dataset
Measure: Number; unit: Participants
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Number analyzed (Participants) | 36 | 27
Participants
  Any Local* | 28 | 23
  Injection site erythema* | 14 | 7
  Injection site induration* | 8 | 5
  Injection site swelling* | 5 | 2
  Injection site warmth* | 4 | 3
  Injection site tenderness* | 23 | 20
  Injection site pain* | 24 | 14
  Any Systemic | 26 | 18
  Chills | 2 | 0
  Malaise | 4 | 3
  Myalgia | 17 | 11
  Arthralgia | 4 | 1
  Headache | 13 | 10
  Fatigue | 13 | 7
  Rash | 2 | 0
  Fever (≥38C) | 0 | 0
  Any Other# | 2 | 2
  Analgesic antipyretic medication used# | 9 | 4
  Stayed at home due to reaction# | 2 | 0

3. Secondary Outcome: The Time Course of HP Infection Following HP Challenge in Vaccinated and Placebo Groups
Description: The time course of HP infection following HP challenge in subjects of the HP vaccine and placebo groups, were assessed by non-invasive HP tests.
Time Frame: 12 months
Measure: Number; unit: Participants
Groups:
- Group I (HP Vaccine): Subjects received three injections of H.pylori(HP) Vaccine at 0, 1, and 2 months, followed by a H.pylori challenge (oral administration of infectious HP inoculum) ≥1 month after 3rd injection.
- Group II (Placebo): Subjects received three injections of Placebo (only aluminum hydroxide adjuvant) at 0, 1, and 2 months, followed by a H.pylori challenge (oral administration of infectious HP inoculum) ≥1 month after 3rd injection.
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Number analyzed (Participants) | 14 | 13
Participants
  Baseline (UBT positive) | 0 | 0
  HP challenge (≥3 months after vaccination) | 0 | 0
  1 week post challenge (UBT positive) | 4 | 1
  2 weeks post challenge (UBT positive) | 1 | 0
  3 weeks post challenge (UBT positive) | 0 | 1
  4 weeks post challenge (UBT positive) | 0 | 1
  8 weeks post challenge (UBT positive) | 0 | 0
  12 weeks post challenge (UBT positive) | 0 | 0
  Post eradication (UBT positive) (N=7,7) | 0 | 0
  Baseline (FAT positive) | 0 | 0
  1 week post challenge (FAT positive) | 9 | 9
  2 weeks post challenge (FAT positive) | 8 | 9
  3 weeks post challenge (FAT positive) | 2 | 5
  4 weeks post challenge (FAT positive) | 3 | 4
  8 weeks post challenge (FAT positive) | 3 | 4
  12 weeks post challenge (FAT positive) | 3 | 1
  Post eradication (FAT positive) (N=7,7) | 0 | 0

4. Secondary Outcome: The Geometric Mean Concentrations After HP Vaccination.
Description: The geometric mean concentration of IgG antibody responses to each of the HP vaccine antigens (VacA, CagA and NAP)after HP vaccination as compared to placebo are reported.
Time Frame: upto 1 month after 3rd vaccination
Population: Per-Protocol dataset
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Number analyzed (Participants) | 35 | 27
μg/mL
  Baseline (CagA antigen) | 2.42 [1.78 to 3.29] | 2.95 [2.09 to 4.18]
  1 month after 1st vaccination (CagA antigen) | 2.89 [1.87 to 4.48] | 2.55 [1.55 to 4.19]
  2 months after 1st vaccination (CagA antigen) | 7.74 [4.83 to 12] | 2.56 [1.5 to 4.39]
  3 months after 1st vaccination (CagA antigen) | 23 [15 to 37] | 2.54 [1.5 to 4.29]
  Baseline (NAP antigen) | 4.59 [3.95 to 5.33] | 5.84 [4.92 to 6.93]
  1 month after 1st vaccination (NAP antigen) | 35 [25 to 50] | 5.47 [3.68 to 8.13]
  2 months after 1st vaccination (NAP antigen) | 236 [175 to 319] | 5.15 [3.66 to 7.24]
  3 months after 1st vaccination (NAP antigen) | 148 [111 to 197] | 2.54 [1.5 to 4.29]
  Baseline (VacA antigen) | 18 [14 to 25] | 21 [15 to 29]
  1 month after 1st vaccination (VacA antigen) | 214 [154 to 298] | 23 [15 to 33]
  2 months after 1st vaccination (VacA antigen) | 2468 [1818 to 3350] | 23 [15 to 33]
  3 months after 1st vaccination (VacA antigen) | 502 [335 to 709] | 19 [13 to 28]

5. Secondary Outcome: Geometric Mean Concentrations Against Vaccine Antigens After HP Challenge.
Description: The geometric mean concentration of IgG antibody responses to each of the HP vaccine antigens (VacA, CagA and NAP) after HP challenge were compared between vaccinated and placebo groups.
Time Frame: 12 months
Population: Per-protocol dataset
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- Group I (HP Vaccine) Infected; Group I (HP Vaccine) Non-Infected: Subjects received three injections of H.pylori(HP) Vaccine at 0, 1, and 2 months, followed by a H.pylori challenge (oral administration of infectious HP inoculum) ≥1 month after 3rd injection.
- Group II (Placebo) Infected; Group II (Placebo) Non-Infected: Subjects received three injections of Placebo (only aluminum hydroxide adjuvant) at 0, 1, and 2 months, followed by a H.pylori challenge (oral administration of infectious HP inoculum) ≥1 month after 3rd injection.
Arm/Group | Group I (HP Vaccine) Infected | Group I (HP Vaccine) Non-Infected | Group II (Placebo) Infected | Group II (Placebo) Non-Infected
Number analyzed (Participants) | 5 | 9 | 6 | 7
μg/mL
  Baseline (CagA) | 2.25 [0.72 to 7.02] | 2.64 [1.13 to 6.16] | 4.17 [1.48 to 12] | 3.53 [1.35 to 9.23]
  1 month after 1st vaccination(CagA ) | 2.24 [0.42 to 12] | 4.54 [1.31 to 16] | 3.84 [0.83 to 18] | 3.06 [0.74 to 13]
  2 months after 1st vaccination (CagA ) | 2.39 [0.51 to 11] | 14 [4.52 to 45] | 4.08 [1 to 17] | 2.95 [0.8 to 11]
  3 months after 1st vaccination (CagA ) | 13 [3.29 to 48] | 93 [34 to 250] | 3.84 [1.13 to 13] | 2.63 [0.85 to 8.12]
  2 weeks post HP challenge (CagA) | 16 [4.39 to 57] | 134 [51 to 348] | 3.92 [1.22 to 13] | 3.59 [1.21 to 11]
  4 weeks post HP challenge (CagA) | 30 [8.89 to 102] | 261 [105 to 648] | 4.11 [1.35 to 13] | 3.39 [1.21 to 9.5]
  12 weeks post HP challenge (CagA) | 149 [35 to 625] | 202 [69 to 588] | 7.51 [2.03 to 28] | 4.73 [1.41 to 16]
  Baseline (NAP) | 4.4 [2.75 to 7.04] | 4.4 [3.1 to 6.24] | 5.46 [3.56 to 8.38] | 11 [7.35 to 16]
  1 month after 1st vaccination (NAP) | 19 [10 to 36] | 62 [39 to 99] | 5.46 [3.11 to 9.59] | 8.48 [5.03 to 14]
  2 month after 1st vaccination (NAP) | 117 [66 to 206] | 235 [154 to 359] | 5.54 [3.3 to 9.31] | 6.61 [4.09 to 11]
  3 month after 1st vaccination (NAP) | 101 [60 to 172] | 251 [170 to 373] | 5.35 [3.3 to 8.66] | 6.59 [4.22 to 10]
  2 weeks post HP challenge (NAP) | 125 [75 to 209] | 275 [187 to 404] | 5.58 [3.49 to 8.49] | 8.3 [5.37 to 13]
  4 weeks post HP challenge (NAP) | 179 [105 to 305] | 325 [219 to 484] | 4.4 [2.7 to 7.16] | 8.32 [5.3 to 13]
  12 weeks post HP challenge (NAP) | 115 [67 to 119] | 208 [139 to 313] | 4.4 [2.68 to 7.24] | 8.01 [5.05 to 13]
  Baseline (VacA) | 21 [9.26 to 47] | 24 [13 to 44] | 20 [9.61 to 42] | 41 [21 to 82]
  1 month after 1st vaccination (VacA) | 117 [46 to 295] | 285 [143 to 569] | 16 [6.89 to 37] | 33 [16 to 70]
  2 months after 1st vaccination (VacA) | 1219 [501 to 2966] | 2754 [1419 to 5344] | 25 [11 to 56] | 33 [16 to 70]
  3 months after 1st vaccination (VacA) | 565 [247 to 1292] | 979 [529 to 1814] | 20 [9.35 to 42] | 34 [17 to 68]
  2 weeks post HP challenge (VacA) | 606 [252 to 1453] | 912 [475 to 1751] | 24 [11 to 53] | 45 [22 to 94]
  4 weeks post HP challenge (VacA) | 2174 [995 to 4752] | 1943 [1085 to 3479] | 28 [14 to 57] | 46 [22 to 94]
  12 weeks post HP challenge (VacA) | 3467 [1632 to 7366] | 1469 [838 to 2577] | 58 [29 to 115] | 73 [39 to 138]

6. Secondary Outcome: Response on Activated Regulatory T Cell Subset Following HP Vaccination and HP Challenge
Description: The response to 3 doses of HP vaccine and the oral HP challenge was assessed with respect their ability to induce differentiation and changes in the phenotype of a subset of regulatory T-cells CD4+CD25+Foxp3+ that expresses Treg Markers PD-1 and/or HLA-DR.
Time Frame: 12 weeks post HP challenge
Population: Per-protocol dataset
Measure: Mean (Standard Deviation); unit: percentage of T-cells
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Number analyzed (Participants) | 19 | 15
percentage of T-cells
  Screening (FOXP3+) | 1.12 (0.33) | 1.13 (0.56)
  HP challenge (FOXP3+) (N=18,15) | 1.15 (0.43) | 1.07 (0.48)
  2 weeks post challenge (FOXP3+) (N=15,14) | 1.34 (0.38) | 1.31 (0.57)
  12 weeks post challenge (FOXP3+)(N=10,9) | 1.34 (0.45) | 0.87 (0.48)
  Screening (HLADR TOT) | 24 (8.22) | 22 (10)
  HP challenge (HLADR TOT) (N=18,15) | 23 (8.36) | 24 (11)
  2 weeks post challenge (HLADR TOT) (N=15,14) | 23 (8.36) | 21 (8.44)
  12 weeks post challenge (HLADR TOT) (N=10,9) | 21 (7.95) | 23 (11)
  Screening (PD-1 TOT) | 5.8 (2.55) | 5.22 (2.06)
  HP challenge (PD-1 TOT) (N=18,15) | 5.69 (1.93) | 5.4 (2.74)
  2 weeks post challenge (PD-1 TOT) (N=15,14) | 6.12 (2.38) | 5.79 (2.52)
  12 weeks post challenge (PD-1 TOT) (N=10,9) | 4.33 (1.31) | 5.53 (2.11)

7. Secondary Outcome: Proliferative Response Against the Pooled H. Pylori Vaccine Antigens by Stimulation Index (SI)
Description: The proliferation of H. pylori-specific Peripheral blood mononuclear cells (PBMCs) following HP antigen stimulation was assessed to measure the magnitude of the cell mediated immune response.
Time Frame: 12 weeks post HP challenge
Population: Per-protocol dataset
Measure: Mean (Standard Deviation); unit: Stimulation Index (SI)
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Number analyzed (Participants) | 20 | 16
Stimulation Index (SI)
  Screening | 6.85 (6.05) | 3.69 (3.7)
  HP challenge (N=21,16) | 26 (21) | 3.81 (2.61)
  2 weeks post challenge (N=17,13) | 53 (37) | 24 (19)
  12 weeks post challenge (N=13,12) | 28 (23) | 7.83 (2.82)

ADVERSE EVENTS:
Time Frame: Throughout the study period (12-14 months)
Arm/Group | Group I (HP Vaccine) | Group II (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/27
Other Adverse Events (participants affected / at risk) | 33/36 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (HP Vaccine) (N=36) | Group II (Placebo) (N=27)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (HP Vaccine) (N=36) | Group II (Placebo) (N=27)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 13 (13) | 7 (7)
Influenza like illness (General disorders) | 8 (8) | 0 (0)
Injection site erythema (General disorders) | 14 (14) | 7 (7)
Injection site induration (General disorders) | 8 (8) | 5 (5)
Injection site pain (General disorders) | 28 (28) | 22 (22)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 5 (5) | 2 (2)
Injection site warmth (General disorders) | 4 (4) | 3 (3)
Malaise (General disorders) | 4 (4) | 3 (3)
Pain (General disorders) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 11 (11)
Headache (Nervous system disorders) | 14 (14) | 10 (10)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days